CLINICAL TRIAL: NCT02528812
Title: Pain Pressure Threshold of a Muscle Tender Spot Increases Following Local and Non-local Rolling Massage
Brief Title: Rolling Massage Decreases Pain Pressure Threshold
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial University of Newfoundland (Other)
Responsible Party: Principal Investigator, Duane Button, Associate Professor, Memorial University of Newfoundland
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 20140537-HK
Record Dates: First submitted 2015-08-14; First posted 2015-08-19 (Estimated); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Manual Lymphatic Drainage

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Ipsi-R (Experimental): Intervention group 1 included participants receiving heavy roller massage via the TheraBand Roller Massager on the calf that exhibited the higher tenderness (Ipsilateral Rolling: Ipsi-R)
  Interventions: Device: TheraBand Roller Massager
- Contra-R (Experimental): Intervention group 2 included participants receiving heavy roller massage via the TheraBand Roller Massager on the calf of the contralateral limb (Contralateral Rolling: Contra-R)
  Interventions: Device: TheraBand Roller Massager
- Sham group (Sham Comparator): The sham group received light stroking of the skin with TheraBand roller massager on the calf that exhibited the higher tenderness
  Interventions: Device: TheraBand Roller Massager
- Ipsi-M (Experimental): Intervention group 3 included participants receiving manual massage on the calf that exhibited the higher tenderness (Ipsilateral Manual: Ipsi-M)
  Interventions: Other: Manual Massage
- control group (No Intervention): received no intervention

INTERVENTIONS:
Device: TheraBand Roller Massager — The roller massager was moved proximal to distal at a slow pace (2 seconds up and 2 second downs) over the muscle belly. Participants in the Sham group received very light pain-free cutaneous strokes of rolling massage with the same pace of rolling as performed for the Ipsi-R and Contra-R groups. The Control group did not receive any treatment.
  Arms: Contra-R; Ipsi-R; Sham group
Other: Manual Massage — A massage therapist massaged the participant
  Arms: Ipsi-M

SUMMARY:
In a randomized control trial and single blinded study, tender spots were identified in 150 participants' plantar flexor muscles (gastrocnemius or soleus). Then participants were randomly assigned to one of five intervention groups (n = 30): 1) heavy rolling massage on the calf that exhibited the higher tenderness (Ipsi-R), 2) heavy rolling massage on the contralateral calf (Contra-R), 3) light stroking of the skin with roller massager on the calf that exhibited the higher tenderness (Sham), 4) manual massage on the calf that exhibited the higher tenderness (Ipsi-M) and 5) no intervention (Control). Pain pressure threshold (PPT) was measured at 30 seconds and up to 15 minutes post-intervention via a pressure algometer.

DETAILED DESCRIPTION:
In a randomized, single blinded, control trial study tender spots were identified in participants' plantar flexor muscles (gastrocnemius or soleus). The acute effect of different roller massage interventions on PPT (i.e. change in PPT from pre- to post-intervention) was investigated. Participants were not informed of the intervention groups. The same registered massage therapist who was blinded to the results of the pre- and post-intervention measurements administered the different modes of massage. In addition, the researcher who recorded the PPT values at pre- and post-intervention levels was blinded to the mode of intervention administered by the massage therapist. It has been shown that the intra-day and inter-day correlations for the algometry muscle tester ranges from 0.88 to 0.99 and 0.94 to 0.98, respectively. The CONSORT guidelines were followed throughout the current research study. The study duration was from June to October 2014.

Experimental protocol. Each participant attended the lab for one experimental session. The participants lay on a massage table in a prone position and a registered massage therapist with more than five years experience examined the relaxed plantar flexor muscles to identify tender spots. A tender spot was identified when an area was hyperirritable on palpation and pressure applied to the area with the pressure pain algometer (with approximately 4 kg/cm2) elicited localized pain greater than 5/10 on a visual analogue scale (VAS). The VAS scale was a horizontal line with anchors at the ends indicating no pain (score of 0) and intolerable pain (score of 10). The identified tender spots were marked with a permanent marker and the spot that exhibited the highest value was chosen for further measurements.

Then the local tenderness (dependent variable) was quantified (by the same massage therapist who screened the participants) measuring the PPT using the pressure pain algometer. The algometer (Lafayette Manual Muscle Test System™, Model 01163, Lafayette Instrument Company, Indiana, USA) was a hand-held muscle tester with a range of 0-300 pounds (136.1 kilograms) that consisted of a padded disc with a surface area of 1.7 cm2 attached to a microprocessor-control unit that measures peak force (pounds or kilograms). The unit has a digital readout for peak-applied pressure and provides a built-in calibration routine that verifies a valid calibration. In order to determine PPT, the researcher would apply the algometer to the tender spot on the participants calf muscle and increase the amount of pressure until the participant verbally informed the researcher when the sensation of pressure became pain at which point the algometer was removed and the PPT value was recorded. PPT values were obtained every 5-10 seconds over the tender spot using a pressure algometer and PPT was measured 6 times. Since the post-intervention PPT measurement was time sensitive, 6 PPT trials with 5-10 seconds interval were performed to gain a consistent value for this measurement.

After completion of pre-intervention PPT measurements, participants were randomly (using a random number generator) assigned to one of five intervention groups. The four massage intervention groups (Ipsi-R, Contra-R, Sham, Ipsi-M) involved 3 sets of 30 seconds massage with 30 seconds of rest between sets. The registered massage therapist performed the roller massage via a Theraband® roller massager (Hygienic Corporation, Akron, OH) technique on the Ipsi-R, Contra-R and Sham groups. The roller massager consisted of a hard rubber material (24 cm in length and 14 cm circumference) with low amplitude, longitudinal grooves surrounding a plastic cylinder. The participants were instructed to provide feedback on the level of perceived pain during the heavy rolling and manual massage (a combination of compressions and petrissage) and the intensity of massage would be adjusted accordingly to ensure 7/10 on the visual analogue scale (VAS) was maintained. The roller massager was moved proximal to distal at a slow pace (2 seconds up and 2 second downs) over the muscle belly. Participants in the Sham group received very light pain-free cutaneous strokes of rolling massage with the same pace of rolling as performed for the Ipsi-R and Contra-R groups. The Control group did not receive any treatment. They lay on the table in prone position for three minutes until post-intervention data was collected. The Control group was assigned in the present study to account for the potential confounding influence of cutaneous touch in Sham.

ELIGIBILITY:
Inclusion Criteria:

* participants had to exhibit point tenderness in their plantar flexor muscles (gastrocnemius or soleus) either in the left or right limb.

Exclusion Criteria:

* having musculoskeletal or visceral chronic pain and taking pain relief medications within the past 24 hours.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2014-04; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Change in Pain Pressure Threshold from pre- to post-interventions | PPT values were obtained over the tender spot and PPT was measured 6 times. PPT measurements were repeated at 2, 5, 10, and 15 minutes following interventions.

CONTACTS AND LOCATIONS:
Overall Officials: Duane Button, PhD, Principal Investigator — Memorial University

REFERENCES:
- [Derived] Aboodarda SJ, Spence AJ, Button DC. Pain pressure threshold of a muscle tender spot increases following local and non-local rolling massage. BMC Musculoskelet Disord. 2015 Sep 28;16:265. doi: 10.1186/s12891-015-0729-5. PMID 26416265